CLINICAL TRIAL: NCT03909022
Title: Assessing Best Medical Treatment Patterns of Patients With Symptomatic Peripheral Arterial Occlusive Disease in Germany - A GermanVasc Study
Brief Title: Assessing Best Medical Treatment Patterns of Patients With Symptomatic Peripheral Arterial Occlusive Disease in Germany
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: GermanVasc (Other); MDEpiNet Chapter Germany (Unknown)
Responsible Party: Principal Investigator, Christian Behrendt, Head of Research Unit GermanVasc and Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: GermanVasc2019_023
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This proposed study will be conducted to support real-world-evidence on the extent of best medical treatment for secondary prevention of patients with symptomatic peripheral arterial occlusive disease (PAOD) for prevention of worsening limb symptoms or of major adverse cardiovascular events. The overall objective of this study is to gain a better understanding of patient characteristics, treatment patterns and outcomes in PAOD patients. For this purpose the investigators will analyze a patient population hospitalized either with intermittent claudication (IC) or chronic limb-threatening ischaemia (CLTI) while taking prior PAOD-related diagnoses in the outpatient setting into account. In detail, we study differentials according to age, calendar time, sex, disease severity and hospital procedure. Data were extracted from available German health insurance claims.

ELIGIBILITY:
1. First clinical diagnosis of symptomatic peripheral arterial occlusive disease (according to Fontaine classification, stages II, III and IV) after at least 5 years without such clinical diagnosis
2. At least 18 years of age

   Exclusion Criteria:
3. Incomplete information on sex, age, date of hospital discharge
4. Less than 5 years of insurance membership before index stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age. Treated in outpatient or inpatient facilities for symptomatic peripheral arterial occlussive disease.
Sampling Method: Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants receiving best-medical-treatment | at 12 months after discharge
  Prevalence of the outpatient prescription of best medical treatment defined as picking up a medication at a pharmacy for a lipid-lowering, an antithrombotic, and an antihypertensive drug agent, within 12 months after index discharge for POAD according to information provided in health insurance claims data

SECONDARY OUTCOMES:
Number of participants deceased | at 5 years after discharge
  Rate of all-cause mortality after index discharge for POAD according to information provided in health insurance claims
Lower extremity amputation | at 5 years after discharge
  Rate of lower extremity amputation after index discharge for POAD according to information provided in health insurance claims
Number of participants with a myocardial infarction | at 5 years after discharge
  Rate of myocardial infarction after index discharge for POAD according to information provided in health insurance claims
Number of participants with a stroke or transient ischaemic attack | at 5 years after discharge
  Rate of stroke or TIA after index discharge for POAD according to information provided in health insurance claims
Number of participants with a major bleeding | at 5 years after discharge
  Rate of major bleeding provided in health insurance claims

CONTACTS AND LOCATIONS:
Overall Officials: Christian-Alexander Behrendt, MD Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Working Group GermanVasc

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peters F, Kreutzburg T, Kuchenbecker J, Debus S, Marschall U, L'Hoest H, Behrendt CA. A retrospective cohort study on the provision and outcomes of pharmacological therapy after revascularisation for peripheral arterial occlusive disease: a study protocol. BMJ Surg Interv Health Technol. 2020 Jan 27;2(1):e000020. doi: 10.1136/bmjsit-2019-000020. eCollection 2020. PMID 35047784
- [Result] Behrendt CA, Sedrakyan A, Peters F, Kreutzburg T, Schermerhorn M, Bertges DJ, Larena-Avellaneda A, L'Hoest H, Kolbel T, Debus ES. Editor's Choice - Long Term Survival after Femoropopliteal Artery Revascularisation with Paclitaxel Coated Devices: A Propensity Score Matched Cohort Analysis. Eur J Vasc Endovasc Surg. 2020 Apr;59(4):587-596. doi: 10.1016/j.ejvs.2019.12.034. Epub 2020 Jan 8. PMID 31926836
- [Result] Peters F, Kreutzburg T, Riess HC, Heidemann F, Marschall U, L'Hoest H, Debus ES, Sedrakyan A, Behrendt CA. Editor's Choice - Optimal Pharmacological Treatment of Symptomatic Peripheral Arterial Occlusive Disease and Evidence of Female Patient Disadvantage: An Analysis of Health Insurance Claims Data. Eur J Vasc Endovasc Surg. 2020 Sep;60(3):421-429. doi: 10.1016/j.ejvs.2020.05.001. Epub 2020 Jul 12. PMID 32669223
- [Derived] Peters F, Kuchenbecker J, Acar L, Marschall U, L'Hoest H, Lareyre F, Spanos K, Behrendt CA. Antithrombotic Treatment Patterns of Patients with Symptomatic Peripheral Arterial Occlusive Disease in Germany: Evidence from Health Insurance Claims Data. J Clin Med. 2022 Sep 16;11(18):5455. doi: 10.3390/jcm11185455. PMID 36143102
- See also: Website of the research group leading this project — http://germanvasc.de